CLINICAL TRIAL: NCT05827328
Title: A Prospective Observational Study to Explore the Optimal Surgical Timing for Lung Surgery and Mediastinal Surgery After COVID-19 Infection
Brief Title: Explore the Optimal Surgical Timing for Lung Surgery and Mediastinal Surgery After COVID-19 Infection
Status: Completed | Type: Observational
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Peng Zhang, Professor, Shanghai Pulmonary Hospital, Shanghai, China
Other Study IDs: COVID-DS
Record Dates: First submitted 2023-04-24; First posted 2023-04-25 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Thoracic Diseases; Thoracic Surgery
MeSH Terms: conditions — Thoracic Diseases | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients eligible for lung surgery or mediastinal surgery: Patients with or without SARS-CoV-2 infection eligible for lung surgery or mediastinal surgery
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Observe the 30-day mortality and 30-day morbidity.

SUMMARY:
Exploring the optimal interval time in patients with the clinical diagnosis of lung cancer or mediastinal tumors indicated for thoracic surgeries after SARS-CoV-2 infection by comparing 30-day mortality and 30-day morbidity.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has fully understood the nature of this study and voluntarily agreed to participate by signing an informed consent form.
2. Participants of any gender between the ages of 18 and 85 are eligible.
3. Preoperative imaging evaluation +/- biopsies indicates that the patient has resectable lung cancer or mediastinal tumors without distant metastasis.

Exclusion Criteria:

1. Patients who have previously undergone lung surgery;
2. Patients previously infected with SARS-CoV-2 more than 6 months before thoracic surgery;
3. Patients who did not receive Chest computed tomography (CT) at admission or within 7 days before surgery, or whose Chest CT at admission suggests pneumonia or current infection with SARS-CoV-2 (confirmed by routine laboratory tests as positive nucleic acid in admission or on the day of surgery);
4. The elapsed time from SARS-CoV-2 diagnosis to surgery is within 4 weeks;
5. Local unresectable lesions or distant metastases are found intraoperatively.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who undergo thoracic surgery for the clinical diagnosis of lung cancer or mediastinal tumors with or without SARS-CoV-2 infection.
Sampling Method: Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2023-01-29 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
The incidence of perioperative mortality | 30 days after surgery
  30-day mortality after surgery

SECONDARY OUTCOMES:
The incidence of perioperative complications | 30 days after surgery
  30-day morbidity after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Peng Zhang, Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China
Locations (6):
- China (6):
  - Shanghai Pulmonary Hospital, Shanghai
  - Anhui Chest Hospital, Shanghai
  - Anqing Municipal Hospital, Shanghai
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai
  - The First Affiliated Hospital of Anhui Medical University, Shanghai
  - Wuhan University Renmin Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No